CLINICAL TRIAL: NCT00742404
Title: A Phase II Study of Pegylated Liposomal Doxorubicin, Bortezomib and Dexamethasone (DVD) for Patients With Newly Diagnosed Multiple Myeloma (MM)
Brief Title: Doxorubicin Hydrochloride Liposome, Bortezomib, and Dexamethasone in Treating Patients With Newly Diagnosed Multiple Myeloma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oncotherapeutics (Industry)
Responsible Party: Regulatory Affairs Associate, Oncotherapeutics
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000612434; ONCOTHER-X05272-DOXILMMY2010; DVD study
Record Dates: First submitted 2008-08-26; First posted 2008-08-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2010-06

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bortezomib; Dexamethasone; Immunologic Techniques

INTERVENTIONS:
Drug: bortezomib
Drug: dexamethasone
Drug: pegylated liposomal doxorubicin hydrochloride
Genetic: protein analysis
Other: immunologic technique

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin hydrochloride liposome and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving bortezomib together with combination chemotherapy may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving doxorubicin hydrochloride liposome together with bortezomib and dexamethasone works in treating patients with newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the response rate (i.e., complete response, very good partial response , partial response, and minimal response) in patients with newly diagnosed multiple myeloma treated with pegylated liposomal doxorubicin hydrochloride, bortezomib, and dexamethasone.

Secondary

* To assess the safety and tolerability of this regimen in these patients.
* To determine the time to disease progression, time to response, duration of response, progression-free survival, and overall survival of patients treated with this regimen.

OUTLINE: Patients receive pegylated liposomal doxorubicin hydrochloride IV over 30-90 minutes, dexamethasone IV, and bortezomib IV on days 1, 4, 8, and 11. Treatment repeats every 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Blood and urine samples are collected at baseline and periodically during study for M-protein analysis by electrophoresis and immunofixation.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma based on the following criteria:

  * Major criteria

    * Plasmacytomas on tissue biopsy (1)
    * Bone marrow plasmacytosis (> 30% plasma cells) (2)
    * Monoclonal immunoglobulin spike on serum electrophoresis IgG > 3.5 g/dL or IgA > 2.0 g/dL and kappa or lambda light chain excretion > 1 g/day on 24-hour urine protein electrophoresis (3)
  * Minor criteria

    * Bone marrow plasmacytosis (10% to 30% plasma cells) (a)
    * Monoclonal immunoglobulin present but of lesser magnitude than given under major criteria (b)
    * Lytic bone lesions (c)
    * Normal IgM < 50 mg/dL, IgA < 100 mg/dL, or IgG < 600 mg/dL (d)
* Meets 1 of the following sets of diagnostic criteria:

  * Any two of the major criteria
  * Major criteria 1 and minor criteria b, c, and d
  * Major criteria 3 and minor criteria a or c
  * Minor criteria a, b, c, OR a, b, d
* Measurable disease, defined as a monoclonal immunoglobulin spike on serum electrophoresis ≥ 1 g/dL and/or urine monoclonal immunoglobulin spike ≥ 200 mg/24 hours, or evidence of lytic bone disease

  * No nonmeasurable disease (i.e., non-secretory or oligosecretory multiple myeloma)
* Symptomatic, newly diagnosed, and previously untreated multiple myeloma
* No POEMS syndrome (i.e., plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein [M-protein], and skin changes)
* No plasma cell leukemia

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Life expectancy > 3 months
* ANC ≥ 1,500/mm^³ (≥ 1,000/mm^³ if bone marrow is extensively infiltrated)
* Platelet count ≥ 75,000/mm^³ (≥ 50,000/mm^³ if bone marrow is extensively infiltrated)
* Hemoglobin ≥ 8.0 g/dL
* AST and ALT ≤ 3.0 times upper limit of normal (ULN)
* Serum bilirubin ≤ 2.0 times ULN
* Creatinine clearance ≥ 30 mL/min OR creatinine > 10 mL/min and < 30 mL/min for patients with significant myelomatous involvement of the kidneys
* Serum potassium ≥ lower limit of normal (LLN)
* Serum sodium ≥ LLN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No peripheral neuropathy ≥ grade 2 within past 14 days
* No impaired cardiac function or clinically significant cardiac disease, including any one of the following:

  * Myocardial infarction within the past 6 months
  * New York Heart Association class II-IV heart failure
  * Uncontrolled angina
  * Clinically significant pericardial disease
  * Severe uncontrolled ventricular arrhythmias
  * LVEF below normal by ECHO or MUGA scan
  * ECG evidence of acute ischemia or active conduction system abnormalities

    * Screening ECG abnormality must be documented by the investigator as not medically relevant
* No severe hypercalcemia (i.e., serum calcium ≥ 14 mg/dL [3.5 mmol/L])
* No poorly controlled hypertension, diabetes mellitus, or other serious medical or psychiatric illness that could preclude study treatment
* No known HIV positivity or hepatitis B or C positivity

  * Baseline testing for HIV and hepatitis B or C is not required
* No history of allergic reaction attributable to compounds of similar chemical or biological composition to doxorubicin, bortezomib, boron, or mannitol

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior or concurrent anti-myeloma therapy except steroids

  * Prior prednisone for ≤ 4 days at a total of 400 mg (or an equivalent potency of another steroid) allowed
  * No concurrent corticosteroids (≥ 10 mg prednisone/day or equivalent) other than dexamethasone
* More than 4 weeks since prior major surgery and recovered

  * Prior kyphoplasty with oncotherapeutic drugs allowed at the investigator's discretion
* More than 4 weeks since prior immunotherapy, antibody therapy, or radiotherapy
* More than 14 days since other prior and no other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Response rate (complete response, very good partial response, partial response, and minimal response) as assessed by modified Bladé criteria at baseline, on day 1 of each course, and at end-of-study

SECONDARY OUTCOMES:
Safety and tolerability as assessed by NCI CTCAE v3.0
Time to progression
Time to response
Duration of response
Progression-free survival
Overall survival
Changes in serum M-protein
Changes in 24-hour urine M-protein

CONTACTS AND LOCATIONS:
Overall Officials: James R. Berenson, MD, Principal Investigator — Oncotherapeutics
Locations (12):
- United States (12):
  - Arizona Clinical Research Center, Incorporated, Tucson, Arizona
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - San Diego Pacific Oncology and Hematology Associates, Incorporated - Escondido, Escondido, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Oncology Care Medical Associates - San Gabriel, Los Angeles, California
  - Desert Cancer Care, Rancho Mirage, California
  - Sutter Cancer Center at Roseville Medical Center, Roseville, California
  - Santa Barbara Hematology Oncology Medical Group at Cancer Center of Santa Barbara, Santa Barbara, California
  - James R. Berenson MD, Incorporated, West Hollywood, California
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - New York Medical College, Valhalla, New York
  - Charleston Hematology Oncology Associates, PA, Charleston, South Carolina